CLINICAL TRIAL: NCT07147829
Title: Digital Silence and Mental Health: The Effects of a Digital Detox Intervention on Depression, Stress, Anxiety, Sleep Quality, and Emotion Regulation in Young Adults: A Randomized Controlled Trial
Brief Title: Digital Silence and Mental Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ceylan Aksoy, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B.30.2.ATA.0.01.00/61811
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Depression Anxiety Disorder; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental)
  Interventions: Behavioral: digital detox

INTERVENTIONS:
Behavioral: digital detox — The digital detox intervention differs from other clinical interventions in several key aspects. Unlike pharmacological treatments or traditional psychotherapy, it focuses on behavioral modification by intentionally reducing or eliminating engagement with digital devices and social media for predetermined periods. The intervention emphasizes mindful technology use, limits screen time, and encourages offline activities to restore emotional balance and improve sleep quality. Additionally, it targets the cumulative effects of constant digital exposure, such as information overload, social comparison, and digital dependency, which are not typically addressed in standard mental health interventions. This unique focus on managing digital behavior positions digital detox as a complementary strategy for promoting psychological well-being in young adults.
  Arms: Intervention Group

SUMMARY:
Social media use has been linked to negative mental health outcomes, including increased anxiety, depression, stress, poor sleep quality, and difficulties in emotion regulation. Digital detox interventions, which involve reducing or temporarily eliminating digital engagement, have emerged as a strategy to mitigate these effects. However, current evidence regarding their effectiveness is mixed and limited by short-term follow-ups and methodological variability. This study aims to examine the impact of a digital detox intervention on depression, anxiety, stress, sleep quality, and emotion regulation in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Owning a smartphone
* Using social media for ≥ 8 hours per day
* Not having a diagnosis related to anxiety, depression, stress, sleep, or emotional regulation
* Living in an environment with internet access
* Providing voluntary informed consent

Exclusion Criteria:

* Having a history of psychiatric diagnosis
* Currently using psychiatric medication
* Having received psychological counseling in the past 6 months
* Having a diagnosis of sleep disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
DASS 21 | 30 day
  The DASS-21 was developed by Lovibond and Lovibond as a shortened version of the DASS-42. The psychometric properties of the Turkish version of the Depression Anxiety Stress-21 (DASS-21) scale in both clinical and non-clinical samples were examined by Sarıçam. In the non-clinical sample, the test-retest correlation coefficients were found to be r = 0.68 for the depression subscale, r = 0.66 for the anxiety subscale, and r = 0.61 for the stress subscale. This scale is a 4-point Likert-type instrument consisting of seven items for each of the three dimensions: depression, anxiety, and stress. A score of 5 or above on the depression subscale, 4 or above on the anxiety subscale, and 8 or above on the stress subscale indicates the presence of the respective problem
PUKİ | 30 day
  The Pittsburgh Sleep Quality Index (PSQI) was developed by Buysse et al. and its validity and reliability in Turkey were established by Ağargün et al. The scale assesses an individual's sleep quality over the past month and consists of 24 items. Nineteen of these are self-report questions, and 18 items are scored across seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each item is rated on a 0-3 scale, with total scores ranging from 0 to 21. Scores of 5 or below indicate "good sleep quality," while scores above 5 indicate "poor sleep quality." The scale demonstrates a high level of internal consistency with a Cronbach's alpha of 0.80, and its diagnostic sensitivity (89.6%) and specificity (86.5%) are also high.

IPD SHARING:
Plan to Share IPD: No